CLINICAL TRIAL: NCT02731898
Title: Fourth International Study of Mechanical Ventilation From VENTILA GROUP
Acronym: ISMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Oscar Penuelas, MD, M.D, Hospital Universitario Getafe
Other Study IDs: ISMV2016
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Failure, Mechanical Ventilation, Critically Ill Patients, Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective, international and multicenter, non interventional single-cohort study, which will enroll consecutive adult patients who have received mechanical ventilation (invasive and noninvasive ventilation) for at least 12 hours during a 1-month period, and will follow each patient for the duration of mechanical ventilation, up to 28 days. The main objectives will be to analyze the mortality and clinical outcomes in ventilated patients and secondly, to evaluate the practices of liberation from mechanical ventilation, the failure of non invasive ventilation in the ICU, and to analyze the clinical outcomes in specific populations of critically ill patients with the need of mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation is commonly used in patients admitted to intensive care units (ICUs). Clinical studies have investigated some of the aspects associated with its utilization, and have contributed to improve the knowledge and management of patients with acute respiratory failure. In 1998, the main researchers conducted the first international study on mechanical ventilation, including 5183 patients who were mechanically ventilated longer than 12 hours. Six years later, the investigators carried out the second international study on mechanical ventilation including 4968 patients. These studies allowed to analyze the evolution of mechanical ventilation and to judge the concordance of practice with results of randomized trials. The main finding of this study was the high degree of concordance between observed changes in mechanical ventilation practice and changes predicted from reports of randomized controlled trials. However, despite apparently beneficial changes in ventilatory practice, the results did not able to detect significant differences in clinical outcomes over this time period. These results have served as an updated benchmark on the usual care and outcomes of mechanically ventilaed patients in a 'real-world' setting. Lastly, in 2010 the main researchers finished the Third International Study of Mechanical Ventilation and were able to find out, for the first time, a significant reduction of ICU mortality in mechanically ventilated patients. Then, the investigators propose to lead up the fourth-international study of mechanical ventilation. This study will keep the same methodology and it will be a prospective, international and multicenter non interventional single-cohort study, which will enroll consecutive patients who have received mechanical ventilation (invasive and noninvasive ventilation) for at least 12 hours during a 1-month period, and will follow each patient for the duration of mechanical ventilation, up to 28 days. Despite of all the current implementations in different ventilatory strategies, and new ventilatory modalities, the mortality and clinical outcomes in critically ill patients under mechanical ventilation is poorly known all over the world. The aims of this study are:

1. To evaluate the impact and clinical outcomes in ventilated patients over the world; and to determine the factors associated with the clinical outcomes in ventilated critically ill patients
2. To analyze the aspects related with the process of liberation from mechanical ventilation;
3. To determine the clinical outcomes of patients with failure of noninvasive ventilation (NIV) in the ICU;
4. To evaluate what differences may occur between geographical areas in the ventilatory management of mechanically ventilated patients.
5. To describe the clinical outcomes in specific populations of critically ill patients with the need of mechanical ventilation:

5.a: Outcomes of prolonged mechanically ventilated patients. 5.b: Prevalence of delirium in mechanically ventilated patients. 5.c: Performance of tracheostomy and outcomes of tracheostomized patients. 5.d: Outcomes of mechanically ventilated patients due to neurologic diseases. 5.f: Outcomes of mechanically ventilated patients due to chronic obstructive pulmonary disease.

5.g: Outcomes of mechanically ventilated patients due to acute renal failure. 5.h: Outcomes of mechanically ventilated patients due to hypercapnia in patients with acute respiratory distress syndrome (ARDS).

5.i: Prediction and Prevalence of ICU acquired weakness (ICUAW) in mechanically ventilated patients.

5.j: Clinical Outcomes and associated factors with reintubation in ventilated patients.

5.k: Clinical Outcomes of elderly patients subjected to mechanical ventilation. 5.l: Clinical impact of the use of sedatives and analgesic drugs in mechanically ventilated patients.

Design of the study This is a multicenter, international, observational and non-interventional study that will collect data of all patients who are admitted to the study ICUs and who meet the inclusion/exclusion criteria between May 1st, 2016 at 00:00 hours and May 31st, 2016 at 23:59 hours. Patients who were already mechanically ventilated prior to April 1 at 00:00 hours will not be included in the study. Approval from the research ethics board of each participating institutions will be sought for this protocol. Only the investigator and research coordinators at each site should be aware of the purpose and the precise timing of the study, in order to minimize any practice modification in response to clinicians' knowledge that they are under observation.

Main variables

For the main purpose of the study we will consider the following variables to fill out:

• Date of ICU admission, mode of mechanical ventilation, date of initiation of mechanical ventilation, demographic dates (age, gender, reason to start mechanical ventilation, severity score at admission, weight, and height), arterial blood gas at the beginning of mechanical ventilation, daily ventilator parameters (applied positive end expiratory pressure [PEEP], volume tidal, peak pressure, plateau pressure), mode of NIV, duration of NIV (failure and success), monitoring during NIV (respiratory rate, sedation scale [Richmond Agitation Sedation Scale, RASS], arterial blood gas during NIV [at the beginning, every 2 hours of NIV if tolerated, and if it failed]), date of the starting of withdrawal of mechanical ventilation, method for weaning in the first attempt, mode of spontaneous breathing trial (SBT), reason for failure of SBT, date of extubation, date of reintubation, arterial blood gas at the time for extubation, reason for reintubation, development of complications during mechanical ventilation (organ failures [cardiovascular, hematological, hepatic or renal failures], barotrauma, ARDS, sepsis, ventilator-associated pneumonia, ICUAW), tracheostomy if needed, date of tracheostomy, type of tracheostomy, date of ICU discharge and status of ICU discharge, reason of ICU mortality, status at hospital discharge, length of ICU and hospital stays.

7. Secondary variables

We consider secondary parameter the following:

• Mode of mechanical ventilation, brand of the ventilator, biochemical parameters during mechanical ventilation, use of co-adjuvant therapies (corticosteroids, insulin therapy), use of medications (neuromuscular blockers, sedatives and analgesics), type of interfaces for NIV, type of respirator for NIV, fluid balance, NIV at home, previous tracheostomy, any isolated ventilator monitoring and setting during mechanical ventilation (invasive or not invasive ventilation), destination after hospital discharge.

STATISTICAL ANALYSIS Randomization This is a prospective, observational, and no intervention study, and therefore, randomization is not applicable.

Sample size calculation Despite of the characteristics of this observational study (an international survey) with multiple objectives to evaluate, we decided to include patients according with the calculation of the sample size for the main objective (ICU mortality). In this way, we estimated that 2,600 patients would need to be enrolled for the study to have 90% power to detect a rate of survival to ICU discharge of 23% versus 28% in the previous study, at an overall two-sided alpha level of 0.05, and assuming 20% of missing patients. The secondary ob-jectives will be tested using the same sample size.

Statistical Methods Appropriate statistical analyses will be conducted. Data will be express as mean (standard deviation), median (interquartile range) and proportion as appropriate. Student's t or Mann Whitney U tests will be use to compare continuous variables and chi-squared tests were used for categorical variables. Statistical analyses will be conducted using appropri-ate statistical software according to evaluated outcome.

Quality Control Extensive efforts will be made to ensure the quality of the data collected throughout the study. At each site, the study physicians, including review of the chart, will review the data from a randomly chosen 5 percent of screened patients and from all patients about whom the screeners had questions. Data from a random sample of 7 percent of cases were abstracted and entered into the database twice, with an error rate of less than 0.25 percent. The charts were reevaluated until the final notes, laboratory test results, and oth-er results will be completed. Complete data will be necessary to include patients in the final analysis, and we will accept patients with no missing data for the main variables or patients with missing data less than 10% for secondary variables.

Ethical and legal issues in this study. Patterns of practices in different hospitals are often idiosyncratic and empiric based in usual care of mechanically ventilated patients.

The study design will provide high quality information about the ventilatory management of critically ill patients from a very large cohort of subjects in a short period of time. It will inform clinical practice much more rapidly than would be possible with a standard randomized clinical trials. Given the study design and the use of anonymous surveys based in routine clinical parameters and ventilatory setting from critically ill patients, the main coordinator team guarantees the ano-nymity of the patients included in the study.

There is no possibility for reporting any adverse events due the type of study (international, pro-spective and non-interventional survey).

Therefore, given the low risk nature of the research (nonintervention study), the anonymity of the survey, and the "unreasonable effort" to get the written informed consent, we will use a pro-cess of "opt-out consent" which involves the provision of information to patients (Information Form) and their next kin and the opportunity to opt-out from the use of their data if they wish.

Confidentiality of patient data Patients will be allocated a unique study code. The site research coordinator will enroll the patient in the international database and the main coordinator of the study will create an enrollment number that include the country, the unit and the unique study code. Study data will be obtained from routinely collected quality assurance. The unique number will identify data entered into the study database only that guarantee the irreversibility of clinical data.

DATA MANAGEMENT Data collection methods All data used in this study are routinely collected from the clinical parameters obtained daily during the ICU admission. These data will be collected by each participating center led by a local coordinator and saved in an online database. This database will be design in the Hospital Universitario de Getafe.

Data monitoring Committee (DMC) A committee of three main investigators (Fernando Frutos Vivar, Óscar Penuelas, Alfonso Muriel) will ensure the rights and safety of patients involved in the study are protected.

FUNDING This study, including the protocol, will be upload in clinicaltrials.com and supported by the Centro de Investigaciones Biomédicas en Red; (CIBER of Respiratory Diseases (CIBER de Enfermedades Respiratorias del Instituto Carlos III) and the Respiratory Group from the Spanish Society of Intensive Care Medicine (Grupo de Respiratorio de la Sociedad Española de Cuidados Intensivos y Unidades Coronarias, SEMICYUC).

This study will not have any financial support. The main researchers of the study does not conflicts of interest to disclosure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are admitted to the ICU and will require invasive mechanical ventilation (endotracheal tube or tracheostomy) longer than 12 hours.
2. Patients who are admitted to the ICU and will require NIV (Continuos Positive Airway Pressure [CPAP], or refers to Bilevel Positive Airway Pressure [BIPAP] with oronasal, nasal, helmet or facial mask) for more than 1 hour.
3. Patients in whom mechanical ventilation was started outside the study ICU at the same Institution and/or a different Institution, including Emergency Room, Operating Room (OR), and were then transferred to the ICU at the participating center.

Exclusion Criteria:

1. Pediatric ICU.
2. Post-Operators Anesthesia Recovery Room.
3. Patients less than 18 years old will be also excluded.
4. Patients admitted after elective surgery and who require mechanical ventilation for less than 12 hours (excepting patients who receive NIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to include patients from different countries and being comparable between them, the coordinator team will create some definitions for the selection of the participating ICUs from each country and inclusion criteria for the patients, as following.
  This study will be conducted in Intensive Care Units ([Medical ICU, MICU], Coronary ICU [CCU], Surgical ICU [SICU], neurocritical ICU) that meet the following criteria:
  1. ICUs that have six or more beds and/or average (during prior 12 months) of more than 30% of the patients admitted requiring mechanical ventilation.
  2. ICUs that have staff specialists in Intensive Care Medicine, or visiting physicians with intensive care training and/or physicians who have more than five years of intensive care experience.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-04-28 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality, | one month
  number of patients admited in the ICU that died during their ICU stay for any cause

SECONDARY OUTCOMES:
duration of mechanical ventilation | one month
  number of days under invasive mechanical ventilation
duration of period of liberation from mechanical ventilation | one month
  number of days from the begining of the period of liberation from mechanical ventilation until the extubation day. In case of tracheostomy, we will considerer the period from the begining of withdrawal from mechanical ventilation until the first 24 hours without ventilatory support
extubation failure | one month
  defined as the need of reintubation within the first 48 hours from a scheduled extubacion
reintubation rate | one month
  number of patients with the need of reintubation, considered by the physician in charge of the patients, after a scheduled or unplanned extubation
tracheostomy rate | one month
  number of patients performed a tracheostomy (either percutaneously or surgical)
28-day mortality | one month
  number of critically ill patients who died within the first 28 days whereever they are (ICU or hospital Ward)
hospital mortality | one month
  number of critically ill patients who died during the hospital admission after the ICU discharge
failure of noninvasive ventilation | one month
  need of orotracheal intubation in critically ill patients after an attempt of noninvasive ventilation that failed, defined by the physician in charge of the patient.
lenght of ICU stay | one month
  period of time that the critically ill patients spend in the ICU and remain discharged (alive or died)
lenght of hospital stay | one month
  period of time that the critically ill patient spend in the hospital after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Penuelas, M.D., Principal Investigator — Hospital Universitario de Getafe, Madrid, Spain
Locations (3):
- Spain (3):
  - Intensive Care Unit, Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Complejo Hospitalario Universitario de A Coruna, A Coruña

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Result] Needham DM, Bronskill SE, Sibbald WJ, Pronovost PJ, Laupacis A. Mechanical ventilation in Ontario, 1992-2000: incidence, survival, and hospital bed utilization of noncardiac surgery adult patients. Crit Care Med. 2004 Jul;32(7):1504-9. doi: 10.1097/01.ccm.0000129972.31533.37. PMID 15241095
- [Result] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] Carlucci A, Richard JC, Wysocki M, Lepage E, Brochard L; SRLF Collaborative Group on Mechanical Ventilation. Noninvasive versus conventional mechanical ventilation. An epidemiologic survey. Am J Respir Crit Care Med. 2001 Mar;163(4):874-80. doi: 10.1164/ajrccm.163.4.2006027. PMID 11282759
- [Result] Schnell D, Timsit JF, Darmon M, Vesin A, Goldgran-Toledano D, Dumenil AS, Garrouste-Orgeas M, Adrie C, Bouadma L, Planquette B, Cohen Y, Schwebel C, Soufir L, Jamali S, Souweine B, Azoulay E. Noninvasive mechanical ventilation in acute respiratory failure: trends in use and outcomes. Intensive Care Med. 2014 Apr;40(4):582-91. doi: 10.1007/s00134-014-3222-y. Epub 2014 Feb 7. PMID 24504643
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Derived] Roca O, Penuelas O, Muriel A, Garcia-de-Acilu M, Laborda C, Sacanell J, Riera J, Raymondos K, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Del Carmen Marin M, Soares MA, Pinheiro BV, Nin N, Maggiore SM, Bersten A, Amin P, Cakar N, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Esteban A, Frutos-Vivar F. Driving Pressure Is a Risk Factor for ARDS in Mechanically Ventilated Subjects Without ARDS. Respir Care. 2021 Oct;66(10):1505-1513. doi: 10.4187/respcare.08587. Epub 2021 Aug 3. PMID 34344717
- [Derived] Mamandipoor B, Frutos-Vivar F, Penuelas O, Rezar R, Raymondos K, Muriel A, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Del Carmen Marin M, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Kelm M, Bruno RR, Amin P, Cakar N, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Wernly B, Esteban A, Jung C, Osmani V. Machine learning predicts mortality based on analysis of ventilation parameters of critically ill patients: multi-centre validation. BMC Med Inform Decis Mak. 2021 May 7;21(1):152. doi: 10.1186/s12911-021-01506-w. PMID 33962603
- [Derived] Wernly B, Bruno RR, Frutos-Vivar F, Penuelas O, Rezar R, Raymondos K, Muriel A, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Marin MDC, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Kelm M, Amin P, Cakar N, Young Suh G, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Guidet B, De Lange DW, Beil M, Svri S, van Heerden V, Flaatten H, Anzueto A, Osmani V, Esteban A, Jung C. Propensity-Adjusted Comparison of Mortality of Elderly Versus Very Elderly Ventilated Patients. Respir Care. 2021 May;66(5):814-821. doi: 10.4187/respcare.08547. Epub 2021 Mar 2. PMID 33653910
- [Derived] Penuelas O, Muriel A, Abraira V, Frutos-Vivar F, Mancebo J, Raymondos K, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Ferguson ND, Del Carmen Marin M, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Amin P, Cakar N, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Esteban A. Inter-country variability over time in the mortality of mechanically ventilated patients. Intensive Care Med. 2020 Mar;46(3):444-453. doi: 10.1007/s00134-019-05867-9. Epub 2020 Jan 7. PMID 31912203
- [Derived] Wernly B, Frutos-Vivar F, Penuelas O, Raymondos K, Muriel A, Du B, Thille AW, Rios F, Gonzalez M, Del-Sorbo L, Del Carmen Marin M, Pinheiro BV, Soares MA, Nin N, Maggiore SM, Bersten A, Kelm M, Amin P, Cakar N, Lichtenauer M, Suh GY, Abroug F, Jibaja M, Matamis D, Zeggwagh AA, Sutherasan Y, Anzueto A, Esteban A, Jung C. Easy prognostic assessment of concomitant organ failure in critically ill patients undergoing mechanical ventilation. Eur J Intern Med. 2019 Dec;70:18-23. doi: 10.1016/j.ejim.2019.09.002. Epub 2019 Oct 9. PMID 31606309